CLINICAL TRIAL: NCT02599181
Title: Local Inflammation Does Not Correlate With Bacterial Colonization and Contamination of Perineural Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNC-Inf
Record Dates: First submitted 2015-09-20; First posted 2015-11-06 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Catheter Infection
Keywords: Perineural cathether; Catheter infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WITH-Group: alcoholic skin disinfection (Experimental): In the WITH-group, the skin is disinfected with an aerosolized alcoholic solution propanol-biphenol: Kodan, Schülke & Mayr, Zurich, Switzerland prior to perineural catheter removal.
  Interventions: Other: propanol-biphenol: Kodan
- WITHOUT: no alcoholic skin desinfection (No Intervention): In the "WITHOUT-group", the skin is NOT disinfected prior to perineural catheter removal.

INTERVENTIONS:
Other: propanol-biphenol: Kodan — WITH-group, the skin is disinfected with an aerosolized alcoholic solutionpropanol-biphenol: Kodan, Schülke & Mayr, Zurich, Switzerland.
  Arms: WITH-Group: alcoholic skin disinfection

SUMMARY:
The aim of this study was to investigate the influence of alcoholic skin disin-fection before PNC (perineural catheter)-removal on the detection of bacteria on the subcutaneous part of the PNC or on the tip. Furthermore, the correlation of bacterial colonization with PNC-associated local inflammation or infection was evaluated.

DETAILED DESCRIPTION:
Two hundred orthopedic patients planned to receive a PNC are prospectively randomized to group PNC-removal with alcoholic skin disinfection or group PNC-removal without skin disinfection.

After standardized PNC-placement under sterile conditions, patients receive a perioperative antibiotic prophylaxis and clinical signs of local inflammation or infection are periodically recorded: The PNC were observed twice daily for clinical signs of local inflammation and local infection. Patients were also evaluated for clinical signs of systemic infection. The adhesive dressing was changed only if it became dislodged or if blood or secretions made visualization of the puncture site impossible. For the dressing change, the anaesthesiologist wore a facemask, a cap and sterile gloves.

Postoperatively, 6 hours after the initial bolus, a local anaesthetic infusion line was connected to the micro filter of the PNC. All patients received patient-controlled perineural analgesia (basal rate 5 ml/h, bolus 4 ml, lock-out time 20 min) with ropivacaine 0.3% for 24 hours, and then reduced to ropivacaine 0.2%.

PNC were removed under sterile conditions after 72h or earlier in the case of signs of infection: Removal of the PNC was performed on the surgical ward by an anaesthesiologist according to a standardized procedure: Wearing a facemask and a cap, the adhesive skin dressing was removed. In the "WITH-group", the skin was now disinfected with an aerosolized alcoholic solution (propanol-biphenol). Procedure continued after three minutes, when the skin was dry with the anaesthesiologist wearing sterile gloves and using sterile tweezers.

The distal part of the PNC (directed to the tip of the PNC) was withdrawn for 1 cm at the insertion site and then cut distally from the tweezers with a sterile pair of scissors. The distal part of the PNC was then totally withdrawn with the sterile tweezers, and with the sterile pair of scissors cut in two parts: the tip (defined as the most distal 2 cm) and the subcutaneous part, which were placed in separate dry sterile containers.

Finally, the remaining proximal part of the PNC was thrown away.

The sterile containers containing the PNC were stored at 4°C and were sent to the laboratory the same day for microbiological analysis of the PNC: The PNC were rolled onto sheep blood agar plates (Becton Dickinson BD, Basel, Switzerland) similar to the semiquantitative culture method for intravenous catheters [10] and thereafter immediately transferred to a liquid enrichment medium (thioglycolate medium, BD Basel Switzerland). Sheep blood agar was incubated for 2 days and thioglycolate for 5 days. In case of growth in the enrichment media only, an aliquot of the liquid was subcultured on solid media. Reports were considered to be positive if any growth was present. Identification of the isolated bacteria and susceptibility testing were performed according to standard methods.

All patients were observed for clinical signs of local infection at the PNC insertion site and for clinical signs of systemic infection one week after PNC-removal. For the correlation of the detection of bacteria on the PNC with clinical signs of in-flammation, the sensitivity, specificity, positive and negative predictive values were calculated on the basis of the following three categories: 1) any growth of bacteria including enrichment, 2) more or equal 5 colonies and 3) more or equal 15 colonies with the semiquantative culture technique, respectively.

ELIGIBILITY:
Inclusion criteria:

Written informed consent, surgery with perineural catheters

Exclusion criteria:

diabetes mellitus, medication with immunosuppressant drugs or any other immune-compromising illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Bacteria detection | After removal of PNC 72h after its insertion
  The reduction of the PNC-colonization rate depending on the removal technique (with or without previous skin disinfection)

SECONDARY OUTCOMES:
sensitivity: to measure the proportion of positives that are correctly identified as such (the percentage of colonized catheters which clinically show an infection). Sensitivity = all clincally positive / all catheters (no unit) | After removal of PNC 72h after its insertion until one week after PNC-removal
  correlation between the Perineural-colonization and clinical signs of local inflammation at the puncture site
Specifity: measures the proportion of negatives that are correctly identified as such (the percentage of not colonized catheters which clinically do not show an infection). Specifity = all clinically negative / all catheters (no unit) | After removal of PNC 72h after its insertion until one week after PNC-removal
  correlation between the Perineural-colonization and clinical signs of local
negative predictive value: all testing negative and no clinical signs of local infection / all testing negative (no unit) | After removal of PNC 72h after its insertion until one week after PNC-removal
  correlation between the Perineural-colonization and clinical signs of local
Positive predictive value: all testing positive and with clinically infection / all testing positive (no unit) | After removal of PNC 72h after its insertion until one week after PNC-removal
  correlation between the Perineural-colonization and clinical signs of local

CONTACTS AND LOCATIONS:
Overall Officials: Alain Borgeat, Prof. MD, Study Director — Balgrist University Hospital, Zurich
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland